CLINICAL TRIAL: NCT00412971
Title: A Randomized, Comparative Phase III, 2-center Study of Hexvix Fluorescence Cystoscopy and Standard Cystoscopy in Patients With Non-invasive Bladder Cancer
Brief Title: A Randomized, Comparative Study of Hexvix Fluorescence Cystoscopy and Standard Cystoscopy in Patients With Non-invasive Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PC B304/04
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer
Keywords: Recurrence of bladder cancer; Fluorescence cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

ARMS (2):
- Hexvix cystoscopy group (Active Comparator)
  Interventions: Drug: Hexvix
- White light (Other): Standard White light cystoscopy
  Interventions: Other: Standard white light cystoscopy

INTERVENTIONS:
Drug: Hexvix — Single installation, TURB
  Arms: Hexvix cystoscopy group
Other: Standard white light cystoscopy
  Arms: White light

SUMMARY:
The main objective of the study is to compare the 1-year recurrence rate of Hexvix assisted Transuretheral Resection of the Bladder (TURB) to standard white light TURB in patients with suspicion of non-invasive bladder cancer.

The hypothesis is to test whether the 1-year recurrence rate is different with Hexvix assisted TURB compared to standard white light TURB.

DETAILED DESCRIPTION:
The main objective of the study is to compare the 1-year recurrence rate of Hexvix assisted Transuretheral Resection of the Bladder (TURB) to standard white light TURB in patients with suspicion of non-invasive bladder cancer.

Patients will be followed 4, 8 and 12 months after the initial TURB. This follow-up regimen is according to standard clinical practice in Denmark.

Recurrence of non-invasive bladder cancer is frequent, and this study is designed to investigate whether Hexvix assisted TURB can reduce the early recurrence compared to standard TURB

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of non-invasive bladder cancer indicated for a transuretheral resection of the bladder
* Above 18 years
* Written informed consent obtained

Exclusion Criteria:

* Gross hematuria. (Note: Gross hematuria is defined as a heavy bladder bleed resulting in marked amounts of blood in the urine, which may interfere with fluorescence cystoscopy. Where the bleed is light, the patient should not be excluded if in the investigator's opinion, rinsing during cystoscopy will alleviate the possible interference with fluorescence cystoscopy).
* Patient with porphyria.
* Known allergy to hexyl aminolevulinate hydrochloride or a similar compound.
* Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days.
* Pregnant or breast-feeding (all women of child-bearing potential must document a negative serum or urine pregnancy test at screening and use the contraceptive pill or intrauterine device (IUD) during the treatments and for at least one month thereafter).
* Conditions associated with a risk of poor protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2005-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregers G Hermann, MD, DM Sci, Principal Investigator — Frederiksberg Hospital
Locations (2):
- Denmark (2):
  - Frederiksberg Hospital, Frederiksberg
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Hermann GG, Mogensen K, Carlsson S, Marcussen N, Duun S. Fluorescence-guided transurethral resection of bladder tumours reduces bladder tumour recurrence due to less residual tumour tissue in Ta/T1 patients: a randomized two-centre study. BJU Int. 2011 Oct;108(8 Pt 2):E297-303. doi: 10.1111/j.1464-410X.2011.10090.x. Epub 2011 Mar 17. PMID 21414125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hexvix Cystoscopy Group | White Light
Started | 115 | 118
Completed | 85 | 108
Not Completed | 30 | 10
Not completed — Lost to Follow-up | 17 | 9
Not completed — Protocol Violation | 13 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hexvix Cystoscopy Group | White Light | Total
Number analyzed (Participants) | 115 | 118 | 233
Age Continuous [Mean (Standard Deviation); unit: years] | 70.6 (11.5) | 69.1 (10) | 69.8 (10.7)
Gender [Number; unit: participants]
  Female | 75 | 81 | 156
  Male | 27 | 36 | 63
Region of Enrollment [Number; unit: participants]
  Denmark | 115 | 118 | 233

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Histologically Confirmed Recurrence Within One 1 Year.
Description: To compare tumour recurrence rates after standard (white light) and fluorescence guided transurethral resection of the bladder (TURB) in patients with macroscopic non-muscle invasive bladder tumour.
Time Frame: 1 year
Population: PP. 145 patients were eligible for tumor recurrence. 12 patients has their last follow up after 12 months. Recurrence after 12 months is based on a total of 133 patients.
Measure: Number (95% Confidence Interval); unit: precentage of participants
Arm/Group | Hexvix Cystoscopy Group | White Light
Number analyzed (Participants) | 59 | 74
precentage of participants | 30.5 [19.2 to 43.9] | 47.3 [35.6 to 59.3]
Statistical Analysis 1: Comparison: Hexvix Cystoscopy Group vs White Light; Test type: Superiority or Other; p = 0.05, Cochran-Mantel-Haenszel; difference in recurrence rate = 0.25

2. Secondary Outcome: Proportion of Patients in the Hexvix Cystoscopy Group Who Had at Least One Additional Lesion Found by Hexvix Cystoscopy That Was Not Found by White Light Cystoscopy.
Time Frame: At day 0
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hexvix Cystoscopy Group
Number analyzed (Participants) | 90
percentage of participants | 48.9 [38.2 to 59.7]

3. Secondary Outcome: False Positive Detection Rate Patient Level
Time Frame: 12 months
Measure: Number; unit: percent of patients
Arm/Group | Hexvix Cystoscopy Group | White Light
Number analyzed (Participants) | 102 | 117
percent of patients | 25 | 16

ADVERSE EVENTS:
Arm/Group | Hexvix Cystoscopy Group | White Light
Serious Adverse Events (participants affected / at risk) | 12/112 | 4/118
Other Adverse Events (participants affected / at risk) | 28/112 | 8/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hexvix Cystoscopy Group (N=112) | White Light (N=118)
Azotaemi (Renal and urinary disorders) | 1 | 0
Oesofageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aortic aneaurysm ruptur (Vascular disorders) | 1 | 0
Phaumonia (Infections and infestations) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 5 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Urinary badder haemorrhage (Renal and urinary disorders) | 0 | 1
Bladder catheter temporary (Surgical and medical procedures) | 0 | 1
Haemutaria (Renal and urinary disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Hypertention (Vascular disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hexvix Cystoscopy Group (N=112) | White Light (N=118)
Urinary retention (Renal and urinary disorders) | 16 | 2
Haematuria (Renal and urinary disorders) | 2 | 3
Bladder perforation (Renal and urinary disorders) | 2 | 1
Cystitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 1
Phyrexia (General disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days